CLINICAL TRIAL: NCT01354574
Title: Thermic & Lipemic Properties of Dietary Carbohydrates
Acronym: FL33
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Nancy L. Keim, USDA, ARS, WHNRC
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 200210295; FL33 (Other: USDA-ARS-WHNRC)
Record Dates: First submitted 2010-08-13; First posted 2011-05-17 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Exogenous Obesity; Dietary Modification
Keywords: energy metabolism; lipids; lipoproteins; satiety; glycemic load; insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Glycemic Index meals (Experimental): Three days of run-in diet with meals containing high glycemic index carbohydrates followed by test day with breakfast meal containing high glycemic index carbohydrates.
  Interventions: Other: High Glycemic Index meals
- Low Glycemic Index meals (Experimental): Three days of run-in diet with meals containing low glycemic index carbohydrates followed by test day with breakfast meal containing low glycemic index carbohydrates.
  Interventions: Other: Low Glycemic Index meals

INTERVENTIONS:
Other: High Glycemic Index meals — Dietary intervention with meals containing high glycemic index carbohydrates. All foods provided to meet the individual's energy needs. Standardized test meal (breakfast)also contained only high glycemic index carbohydrates and energy content was adjusted for each individual, providing 40% of daily energy needs.
  Other Names: Low Fiber Meals
  Arms: High Glycemic Index meals
Other: Low Glycemic Index meals — Dietary intervention with meals containing low glycemic index carbohydrates. All foods provided to meet the individual's energy needs. Standardized test meal (breakfast)also contained only low glycemic index carbohydrates and energy content was adjusted for each individual, providing 40% of daily energy needs.
  Other Names: High fiber meals
  Arms: Low Glycemic Index meals

SUMMARY:
The purpose of this study is to determine if consumption of meals containing carbohydrates with different glycemic index (a high glycemic index meal and a low glycemic index meal)have different effects on energy expenditure, type of metabolic fuels used for energy, blood lipids and lipoproteins, and sensations of hunger, fullness, and the hormones related to satiety.

DETAILED DESCRIPTION:
Little is known about the metabolic effects of chronic dieting and weight cycling in humans, but limited evidence suggests that fatty acid oxidation may be depressed leading to periodic elevation of circulating lipids associated with meal ingestion and preferential storage of fat in adipose tissue. With the traditional approach of restrictive dieting failing to result in permanent weight loss and, possibly producing abnormalities in lipid metabolism, it is important to evaluate alternative approaches to achieve a healthy body weight through improved metabolism. In this study the investigators will test the postprandial metabolic effects of standard mixed meals containing carbohydrates with high glycemic index and compare these effects to responses obtained with standard mixed meals, matched for protein and fat content but containing carbohydrates with low glycemic index.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 25 and 30 kg/m2
* Having regular menses
* Willing to refrain from restrictive dieting during the course of the study

Exclusion Criteria:

* Pregnant or currently planning a pregnancy
* Cigarette smoking
* Taking medications to induce weight loss or change appetite
* History of cardiovascular disease
* History of metabolic disorders, including diabetes

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Gas Exchange | 30 minutes before a standardized test meal and intermittently for 480 minutes following the meal.
  Respiratory Gas Exchange will be measured using an automated metabolic cart. Gas analyzers and volumeter will be calibrated using manufacturer's procedures.

SECONDARY OUTCOMES:
Plasma glucose | 10 blood samples taken over a 480 minute period.
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of standardized test meal.
Circulating lipoproteins | 4 blood samples taken over a 480 minute period
  Blood samples for lipoprotein analyses were taken at fasting (0 minute) and at 150, 210, and 480 minutes following consumption of test meal. A subset of 10 randomly-selected subjects was chosen for this outcome measure
Subjective evaluation of appetite | 16 timepoints measured over 600 minutes
  Visual analog scales were used to assess appetite-related sensations. Four responses were obtained during the fasting phase (120 minutes) and 12 responses were obtained in the 480 minute postprandial period.
Food consumption at a buffet-style meal | at 480 minutes following test meal
  The amount and types of foods consumed were measured after subject was presented with a buffet-style meal.
Body composition | measured the morning of the standard meal challenge
  Body composition (fat mass, % fat, lean mass, bone density) will be measured using dual energy x-ray absorptiometry.
Serum insulin | 10 blood samples taken over a 480 minute time period
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of test meal.
Plasma leptin | 10 blood samples taken over a 480 minute period
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of test meal.
Plasma ghrelin | 10 blood samples taken over a 480 minute time period
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of test meal.
Cholecystokinin (CCK) | 10 blood samples taken over a 480 minute time period
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of test meal.
GLP-1 | 10 blood samples taken over a 480 minute time period
  1 fasting blood sample (0 minutes) and 9 post-prandial blood samples taken at 30, 60, 90, 120, 150, 210, 270, 360 and 480 minutes following consumption of test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Keim, PhD, Principal Investigator — USDA, ARS, WHNRC
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Result] Motton DD, Keim NL, Tenorio FA, Horn WF, Rutledge JC. Postprandial monocyte activation in response to meals with high and low glycemic loads in overweight women. Am J Clin Nutr. 2007 Jan;85(1):60-5. doi: 10.1093/ajcn/85.1.60. PMID 17209178
- [Result] Burton-Freeman BM, Keim NL. Glycemic index, cholecystokinin, satiety and disinhibition: is there an unappreciated paradox for overweight women? Int J Obes (Lond). 2008 Nov;32(11):1647-54. doi: 10.1038/ijo.2008.159. Epub 2008 Sep 30. PMID 18825157